CLINICAL TRIAL: NCT04436783
Title: Virtual Reality Epley Maneuver System (VREMS) for Treatment of Benign Paroxysmal Positional Vertigo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Euna Hwang, Otolaryngologist, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REB19-1367
Record Dates: First submitted 2020-05-26; First posted 2020-06-18 (Actual); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: BPPV; Vertigo, Peripheral
Keywords: BPPV; Vertigo; Peripheral vestibular disorder; Virtual reality
MeSH Terms: conditions — Vertigo

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Epley Maneuver System - VREMS (Experimental): Patients in the VREMS cohort will be provided with the VREMS device, which will help guide them through the Epley maneuver in a virtual reality environment. All participants will be asked to rate the severity of their symptoms before undergoing the Epley maneuver. Subsequently, patients will be supervised as they perform the Epley maneuver - VREMS assisted. In both groups, once the patient has performed the Epley maneuver (whether with VREMS assistance or with the IH), they will be asked to rate their symptom severity after undergoing the Epley maneuver
  Interventions: Device: Virtual Reality Epley Maneuver System (VREMS)
- Instructional Handout (IH) (Active Comparator): Those in the control cohort will be provided an instructional handout (IH) to help them perform the Epley maneuver. They will be given a chance to review the IH, and then they will have a chance to perform the Epley maneuver.
  Interventions: Other: Instructional Handout (IH)

INTERVENTIONS:
Device: Virtual Reality Epley Maneuver System (VREMS) — The VREMS system includes a smartphone placed inside virtual reality goggles worn by the participant. On the smartphone there is a virtual reality application. When viewed through the VR goggles the participants see a three-dimensional environment. Audio and text cues are presented in a 3D environment to help guide the patient through the Epley maneuver.
  Arms: Virtual Reality Epley Maneuver System - VREMS
Other: Instructional Handout (IH) — Patients randomized to the IH group will be given an instructional handout with image and text-based instructions on the steps involved in performing the Epley maneuver. They will then be given the chance to perform the Epley maneuver.
  Arms: Instructional Handout (IH)

SUMMARY:
Background and Rationale:

Benign paroxysmal positional vertigo (BPPV) is the most common cause of vertigo, affecting 2.4% of the general population and 30% of those over 70 years old. The main symptom is the perceived sensation of movement of the surrounding or self, without actual such movement, triggered by changes in position (positional vertigo). It can be dangerous as repetitive symptoms can lead to falls and depression, particularly in the elderly. Additionally, at least half of those with initial symptoms of BPPV will have ongoing symptoms if not treated. The Epley maneuver is a particle-repositioning maneuver that is used to treat posterior semicircular canal BPPV, the most common type of BPPV, after a diagnosis has been made on physical examination. In-office administration of the Epley maneuver by a specialist yields a 90% success rate at treating the condition; however, at-home administration is much less successful. In a previous paper we demonstrated the development and face validation of a Virtual Reality Epley Maneuver System (VREMS) for performing the Epley maneuver correctly. In this study we aim to apply VREMS treatment in patients who have been diagnosed with BPPV.

Research Question and Objectives:

PICO (Patient/Population Intervention Compare Outcome): In adult patients diagnosed with posterior canal BPPV by a specialist, does VREMS, as compared to self-performed Epley maneuver using an instructional handout (IH) result in improved or resolved symptoms?

Methods:

Vertigo patients referred to the Neurovestibular Clinic will be evaluated by an Ear, Nose and Throat (ENT) specialist. Those who are diagnosed with posterior canal BPPV after history and physical examination including the Dix-Hallpike test will be approached to be recruited into the study. Patients who consent to participating in the study will be allocated to either the VREMS cohort or the control cohort. Those in the control cohort will be provided an instructional handout (IH) to help them perform the Epley maneuver. Patients in the VREMS cohort will be provided with the VREMS device, which will help guide them through the Epley maneuver in a virtual reality environment. All participants will be asked to rate the severity of their symptoms before undergoing the Epley maneuver. Subsequently, patients will be supervised as they perform the Epley maneuver - VREMS assisted or based on reading the IH. In both groups, once the patient has performed the Epley maneuver (whether with VREMS assistance or with the IH), they will be asked to rate their symptom severity after undergoing the Epley maneuver. All patients will also be asked to complete the NASA Task Load Index (NASA-TLX) to gauge their perceived mental workload. They will also be given an opportunity to give free-text feedback. For any patient with residual BPPV symptoms following Epley maneuver with VREMS or IH, the ENT specialist/vestibular physiotherapist will perform the Epley maneuver to ensure resolution of symptoms if possible prior to discharge from the clinic. The primary outcome of the study will be the improvement in and resolution of BPPV symptoms with VREMS use as compared to IH. Secondary outcome will be mental workload in each of the study arms.

ELIGIBILITY:
Inclusion Criteria:

* Adults (over 18 years old)
* Clinical diagnosis of posterior semicircular canal benign paroxysmal positional vertigo

Exclusion Criteria:

* Hemodynamically unstable
* Cervical spine instability
* Limited neck range of motion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-11-14 (Estimated); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Subjective dizziness | Self reported once immediately before performing the Epley maneuver and once immediately after - in both arms
  Patient reported dizziness score out of 10 - Min value 0(no dizziness) and max value 10 (completely debilitating dizziness). The higher the score, the greater the subjective dizziness (worse outcome).

SECONDARY OUTCOMES:
Mental demand | Reported once immediately before performing the Epley maneuver and once immediately after - in both arms
  Mental demand reported using the National Aeronautics and Space Administration (NASA) - Task Load Index - Minimum score 0 (no mental demand) and maximum score is 100 (very high mental demand). The higher the score, the greater the mental demand (worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Euna Hwang, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hanley K, O'Dowd T, Considine N. A systematic review of vertigo in primary care. Br J Gen Pract. 2001 Aug;51(469):666-71. PMID 11510399
- [Background] Kuo CH, Pang L, Chang R. Vertigo - part 1 - assessment in general practice. Aust Fam Physician. 2008 May;37(5):341-7. PMID 18464964
- [Background] Strupp M, Brandt T. Diagnosis and treatment of vertigo and dizziness. Dtsch Arztebl Int. 2008 Mar;105(10):173-80. doi: 10.3238/arztebl.2008.0173. Epub 2008 Mar 7. PMID 19629221
- [Background] von Brevern M, Radtke A, Lezius F, Feldmann M, Ziese T, Lempert T, Neuhauser H. Epidemiology of benign paroxysmal positional vertigo: a population based study. J Neurol Neurosurg Psychiatry. 2007 Jul;78(7):710-5. doi: 10.1136/jnnp.2006.100420. Epub 2006 Nov 29. PMID 17135456
- [Background] Hall SF, Ruby RR, McClure JA. The mechanics of benign paroxysmal vertigo. J Otolaryngol. 1979 Apr;8(2):151-8. PMID 430582
- [Background] Gopinath B, McMahon CM, Rochtchina E, Mitchell P. Dizziness and vertigo in an older population: the Blue Mountains prospective cross-sectional study. Clin Otolaryngol. 2009 Dec;34(6):552-6. doi: 10.1111/j.1749-4486.2009.02025.x. PMID 20070765
- [Background] Neuhauser HK, Radtke A, von Brevern M, Lezius F, Feldmann M, Lempert T. Burden of dizziness and vertigo in the community. Arch Intern Med. 2008 Oct 27;168(19):2118-24. doi: 10.1001/archinte.168.19.2118. PMID 18955641